CLINICAL TRIAL: NCT07012746
Title: A Randomized, Double-Blind, Placebo-Parallel-Controlled Clinical Trial to Explore the Safety and Efficacy of TJ0113 Capsules in the Treatment of Patients With Age-related Hearing Loss
Brief Title: A Clinical Trial of the Safety and Efficacy of TJ0113 Capsules in the Treatment of Patients With Age-related Hearing Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yilai Shu (Other)
Collaborators: Hangzhou PhecdaMed Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yilai Shu, Principal Investigator, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024198-1
Record Dates: First submitted 2025-04-29; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Age Related Hearing Loss; Deafness
MeSH Terms: conditions — Presbycusis; Deafness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TJ0113 group (Experimental): Participants will be treated with TJ0113 capsule 200 mg daily for up to 24 weeks
  Interventions: Drug: TJ0113 capsules
- Placebo group (Placebo Comparator): Participants will be treated with a placebo 200 mg daily for up to 24 weeks
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: TJ0113 capsules — Oral intake on an empty stomach in the morning, 200 mg each time, fasting within half an hour after taking. It is recommended to keep the drug at the same time (± 1 h ) of a day .
  Arms: TJ0113 group
Drug: Placebo capsules — Oral intake on an empty stomach in the morning, 200 mg each time, fasting within half an hour after taking. It is recommended to keep the drug at the same time (± 1 h ) of a day .
  Arms: Placebo group

SUMMARY:
The purpose of this study is to explore the safety and efficacy of TJ0113 capsules in patients with age-related hearing loss.

DETAILED DESCRIPTION:
The main purpose of this clinical trial is to explore the safety of TJ0113 capsules in patients with age-related hearing loss; the secondary purpose is to explore the effectiveness; and the exploratory purpose is to exploring changes in muscle strength, depression degree, cognition, and biomarkers after TJ0113 capsule treatment in patients with age-related hearing loss. Approximately 60 subjects (aged from 65~75) will be enrolled in this study according to the randomization and drug randomization tables both of which were generated by computer. The successfully screened subjects were randomly assigned to the 1:1 TJ0113 capsule group (n=30) and placebo group (n=30).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participate in the clinical trial, sign the informed consent form, understand and follow the protocol, and fully understand the test content, process and possible adverse reactions.
2. Age between 65 and 80 years (including the critical value)
3. A diagnosis of symmetrical sensorineural deafness (SNHL) with a history of> 3 months (binaural threshold difference in mean PTA frequency <15 dB HL), the PTA level should be between moderate (> 35dB) and severe (<80dB) hearing loss
4. Hearing aids have not been used, or otherwise, it should be used regularly for more than 3 years and stopped for 3 months before enrollment.
5. Subjects and their partners had no birth plan, sperm or egg donation plans from the screening period until within 6 months after the end of the trial and would voluntarily take effective contraception (e. g. abstinence, condoms, etc.). Male subjects should agree to avoid sperm donation within 6 months from the start of administration until cessation of study treatment. Female subjects should be menopausal (over 24 months).

Exclusion Criteria:

1. The presence of implants in the study ear (such as cochlear implant, artificial hearing bone, etc.);
2. Suffering from acute otitis media or other ear infection within the previous 3 months or previous chronic suppurative otitis media or tympanic membrane perforation, or with conductive deafness, previous history of ear trauma or surgery, combined middle ear or inner ear malformation, otosclerosis, Meniere's disease, sudden deafness and no recovery of hearing, all of which will impact results explained.
3. Patients with sensorineural deafness caused by non-aging factors (e. g., hereditary deafness, congenital deafness, drug-induced deafness, noise deafness, neurosyphilis, severe retrocochlear lesions or organic lesions), and unilateral deafness
4. Occupation that is sensitive to sound: musician, conductor, music teacher, etc.
5. Use headphones at high volume or frequent exposure to noise in previous work or life;
6. History of alcohol or drug dependence / drug abuse in the last 1 year;
7. Positive pregnancy test at screening or at the baseline visit, pregnant, lactating, or planned to become pregnant during the trial

7.Failure to swallow oral medication, or, according to the investigator, any conditions that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or that may pose a hazard to the subjects participating in this trial; 9.People who currently taking drugs that can improve symptoms such as dementia and depression 10.Subjects with a severe or unstable systemic disease, such as serious congenital disease, blood disease, endocrine disease, nerve or nervous system disease, end-stage disease, head and neck tumor radiotherapy and chemotherapy history, major surgical treatment, psychological disorders (severe insomnia, severe depression, severe anxiety, etc. diagnosed within the previous 90 days ) or history and clinical significance of abnormal baseline laboratory values, such as hepatic insufficiency (alanine transaminase (ALT) and / or alanine transaminase (AST) is 2 times above the upper limit of the reference range, or renal insufficiency (creatinine clearance Ccr <30 mL/min), or history of malignant tumors and the detection results of tumor markers during the screening period have clinical significance, or unsuitable participants, as judged by the investigator; 11.Subjects suffering from any one of the following heart diseases: a. having uncontrolled or serious cardiovascular and cerebrovascular disease, including the development of grade II ( New York Heart Association, NYHA) or above congestive heart failure, unstable angina, acute myocardial infarction within 6 months before the first drug administration, or cardiac arrhythmias requiring treatment at screening; With b. hypertension (systolic pressure≥ 160mmHg and / or diastolic v≥ 100mmHg), and after the combination of two or more antihypertensive drugs can not be reduced to the normal range; or c.with a history of clinically significant ECG abnormalities, the QRS time was> 120ms, Long QT syndrome: QTc interval> 450ms in male or QTc interval> 470ms in female.

12.Participated in a clinical study involving the administration, device, or surgery of the study drug (new chemical entity) within 90 days or 5 half-lives (whichever is longer) 13.Patients with a previous history of hepatitis B, or any of the following indicators are positive at screening: hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody.

14.The subject is not fit to participate in the study if the investigator considers. Or the subject could not participate in the trial for his own reasons, or the behavior subject may interfere with treatment, study or interpretation of results (e. g., previous treatment with high-dose aminoglycosides).

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety of TJ0113 capsule in the treatment of patients with age-related hearing loss | Baseline, weeks 1, 4, 12, 24, and 1 week after discontinuation
  Incidence of adverse events in each group

SECONDARY OUTCOMES:
Speech Intelligibility - Word Recognition in Quiet and Noise | From baseline to 4, 12 ,24 weeks
  To compare the change in word list-measured recognition accuracy rates for words and short sentences in both quiet and noise.
Pure Tone Audiometry (PTA) | From baseline to 4, 12 ,24 weeks
  To ompare the change in Pure Tone Audiometry (PTA) using the air and bone conduction audiometry for hearing at certain range (Hz).
Individual's health-related quality of life (HRQOL) | From baseline to 4, 12 ,24 weeks
  SF-36 quality of life questionnaire will be measured to compare the change in individual's health-related quality of life using face to face Interview for the scores. Higher scores mean better functioning or fewer symptoms.

OTHER OUTCOMES:
Auditory brainstem response (ABR) | From baseline to 12 and 24 weeks
  To compare the change in the auditory brainstem response (ABR) using the threshold (dB). Higher thresholds indicate worse outcomes.
Distortion product otoacoustic emissions (DPOAE) | From baseline to 12 and 24 weeks
  To compare the changes in the pass rate levels of distortion product otoacoustic emissions（DPOAE).
Tinnitus Assessment | From baseline to 4, 12 and 24 weeks
  Tinnitus Handicap Inventory (THI) questionnaire scores will be measrued to compare the change in tinnitus using face to face Interview for the scores. Higher scores indicate worse outcomes.
Muscle strength | From baseline to 4, 12 and 24 weeks
  To compare the change in the muscle strength (kg) measured with a handgrip dynamometer.
Depression levels | From baseline to 4, 12 and 24 weeks
  To compare the change in depression levels using face to face Interview for the Geriatric depression scale-15 (GDS-15) scores.
Cognition | From baseline to 4, 12 and 24 weeks
  To compare the change in cognition by Montreal cognitive gssessment (MoCA) using face to face Interview for the scores.
Plasma Senescence-associated secretory factor (SASP) | From baseline to 24 weeks
  The absolute values of changes in the levels of plasma Senescence-associated secretory factor (SASP) related to the mechanism. The concentration of the plasma Senescence-associated secretory factor will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No